CLINICAL TRIAL: NCT05400018
Title: Clinical Evaluation of Genetron D842V PCR Kit in GIST Patients
Status: Completed | Type: Observational
Sponsor: Genetron Health (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other); Harbin Medical University (Other); Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20200196
Record Dates: First submitted 2022-05-23; First posted 2022-06-01 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: GIST; Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this trail is to evaluate the performance of Genetron D842V PCR kit in GIST patients using real-time PCR method.

DETAILED DESCRIPTION:
This trial follows the principle of synchronous blinding. The enrolled cases are coded, and the enrolled samples are detected with Genetron D842V PCR Kit and Sanger sequencing method. The results were determined independently according to the cutoff values or interpretation requirements provided by each method. The safety and effectiveness of this kit are confirmed and evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Paraffin-embedded tissue samples from patients clinically diagnosed with gastrointestinal stromal tumor (GIST), and a small number of other cancers or benign lesions in the gastrointestinal site were included as interference samples.
2. The sample should have corresponding basic clinical information, including: the patient's unique traceability number, age, gender, pathological diagnosis results, etc.
3. The sample is a formalin-fixed paraffin-embedded gastrointestinal stromal tumor tissue sample, and each sample can provide 5 paraffin sections or 5 paraffin rolls with a thickness of at least 5 µm.
4. The content of tumor cells meets the requirements of assessment reagents and comparison methods.

Exclusion Criteria:

1. The investigator considers that it is not appropriate to continue the clinical trial, such as the samples that are not prepared according to the required steps.
2. Samples that cannot complete the entire testing process.
3. Patients with incomplete sample information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital sample
Sampling Method: Non-Probability Sample
Enrollment: 1041 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Ct Value (Ct Values From PCR Reaction) | 3 months
  the number of PCR cycles where the amplification signal starts to be observed

SECONDARY OUTCOMES:
PPV | 3 months
  the ratio of true positive in all positive cases
NPV | 3 months
  the ratio of true negative in all negative cases
Consistency (the Overall Ratio of True Positive and True Negative) | 3 months
  The overall consistency ratio of true positive and true negative, i.e. (true positive+true negative)/total number of cases
Kappa coefficient | 3 months
  Kappa coefficient is the consistency analysis of the extent of agreement between the test results of the Genetron D842V PCR kit and sanger sequencing method.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking University Cancer Hospital, Beijing
  - Harbin Medical University Cancer Hospital, Harbin
  - Shanghai Tenth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT05400018/Prot_000.pdf